CLINICAL TRIAL: NCT05036811
Title: HIV and Inflammatory or Autoimmune Disease: Rare Patients, Many Questions (MAIVIH)
Acronym: MAIVIH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NRIPH_2020_11
Record Dates: First submitted 2021-04-16; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-04

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection — data collection

SUMMARY:
Follow-up registry of patients living with HIV who also have various inflammatory and autoimmune pathologies that may require immunosuppressive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient living with HIV
* Carrier of one or more of the following diseases:

Sarcoidosis Multiple sclerosis Myasthenia gravis Crohn's disease Hemorrhagic rectocolitis Autoimmune hepatitis Arthropathic psoriasis Still's disease, other rheumatoid arthritides, juvenile polyarthritides, Rheumatoid arthritis Vasculitides: periarteritis nodosa and related conditions, other necrotizing vasculopathies (periarteritis nodosa, juvenile periarteritis, Churg-Strauss disease, polyangiitis, Kawasaki disease, Horton's disease, Wegener's disease, thrombotic microangiopathy, Takayashu syndrome, Good-Pasture's syndrome, thrombocytopenic purpura) Lupus Polymyositis or dermatopolymyositis Connectivitis (Behcet's disease, Gougerot-Sjöogren syndrome) Inflammatory spondyloarthropathies (APS, spondyloarthritis, other spondyloarthropathies)

Exclusion Criteria:

* Opposition of the person
* Minor patients
* Patients under judicial protection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with HIV and an inflammatory or autoimmune disease
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients living with HIV who have an inflammatory or autoimmune disease | At the end of the study an average of 18 months

SECONDARY OUTCOMES:
Number of patients on immunosuppressive treatment, | At the end of the study an average of 18 months
Occurrence of infectious complications | At the end of the study an average of 18 months
Number of patients on remission | At the end of the study an average of 18 months
Evolution of CD4 and HIV viral load | At the end of the study an average of 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie VIGET, MD, Principal Investigator — CH TOURCOING
Locations (1):
- CH Tourcoing, Tourcoing, France

IPD SHARING:
Plan to Share IPD: No